CLINICAL TRIAL: NCT00804115
Title: The International Collaborative Exfoliation Syndrome Treatment Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The New York Eye & Ear Infirmary (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Robert Ritch, MD, Glaucoma Associates of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00.24
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Exfoliation Syndrome; Glaucoma; Ocular Hypertension
Keywords: Exfoliation Syndrome; Latanoprost; Timolol; Pilocarpine
MeSH Terms: conditions — Exfoliation Syndrome; Glaucoma; Ocular Hypertension | interventions — Latanoprost; dorzolamide-timolol combination; Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Latanoprost in combination with Pilocarpine
  Interventions: Drug: Latanoprost with Pilocarpine vs Timolol or Cosopt
- 2 (No Intervention): Timolol or Cosopt
  Interventions: Drug: Latanoprost with Pilocarpine vs Timolol or Cosopt

INTERVENTIONS:
Drug: Latanoprost with Pilocarpine vs Timolol or Cosopt — Timolol 0.5% bid or Cosopt bid Latanoprost 0.005% qhs Pilocarpine 2%
  Other Names: Timolol; Cosopt

SUMMARY:
Purpose: To determine the efficacy of treatment with latanoprost in combination with pilocarpine versus timolol or timolol/dorzolamide fixed combination (Timoptic or Cosopt) in eyes with XFS and elevated intraocular pressure (IOP).

Methods: This is a randomized, open-label study to test the hypothesis that improving both pressure-dependent and pressure-independent aqueous outflow and minimizing iridolenticular friction will interfere with the progression of XFS, allow improvement in trabecular function, and be more effective over time than simply reducing aqueous formation. Randomization was performed across the centers, per patient rather than per eye to avoid any crossover effect caused by aqueous suppressants. Group I was treated with latanoprost and pilocarpine, both in the evening, and Group II with Timolol or Cosopt b.i.d. Only one eye per patient was randomized. Patients were followed for 2 years with assessment of IOP, visual field progression, tonographic outflow coefficient and trabecular pigmentation at the 6:00 and 12:00 position.

DETAILED DESCRIPTION:
Purpose: To compare the effect of treatment with latanoprost plus pilocarpine vs timolol or fixed combination timolol/dorzolamide (T/D) in eyes with exfoliation syndrome (XFS) and elevated IOP.

Methods: A randomized, prospective, international, 12-center, two-year, open-label clinical trial was conducted. XFS patients aged 50-80 years with untreated IOP ≥22 mmHg and open angles with or without mild to moderate glaucomatous damage were included. One eligible eye per patient was randomly assigned to latanoprost and pilocarpine qhs to increase aqueous outflow and inhibit pupillary movement (group I), or to decrease aqueous production with timolol or T/D bid as needed for IOP control (group II). IOP, tonographic outflow facility, and trabecular pigmentation were measured every 6 months.

Results: 277 (146 male) patients (mean age 69.1±6.8 yr, range 50-80 yr)' were enrolled between October 2000 and July 2003. XFS was unilateral in 118 (42.6%) and bilateral in 159 (57.4%) patients. Baseline TM pigmentation at the 6:00 angle was significantly associated with IOP (p=0.01). IOP reduction was 1.3 mmHg greater in Group I (n=145) than in Group II (n=132) (p=0.0003). Mean increase in outflow facility in Group I was 0.005 µl/mmHg/min vs 0 μl/mmHg/min in Group II (p<0.001). TM pigmentation at the 6:00 position at 24 months decreased from baseline more frequently in Group I than in Group II [34(26%) vs 20(16%)] and increased from baseline more frequently in Group II than in Group I [31(25%) vs 24(18%)].

Conclusions: Subjects in Group I had lower IOP, improved outflow facility and decreased TM pigmentation. Initial therapy to increase aqueous outflow and interfere with dispersion of exfoliation material and iris pigment by inhibiting pupillary movement is preferable to reducing aqueous secretion, which may be deleterious as primary treatment in this disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Exfoliation syndrome in one or both eyes. Exfoliation material must be present on the anterior lens surface for diagnosis.
2. Untreated IOP greater than or equal to 22 mmHg in one or both eyes with or without mild to moderate glaucomatous damage and who, in the judgment of the investigator, can be safely washed off from current medical therapy.
3. Age 50-80 years
4. Open angles by gonioscopy

Exclusion Criteria:

1. Age over 80 years
2. Best corrected visual acuity less than 20/30
3. Untreated IOP greater than 35 mmHg
4. Currently taking systemic beta-blockers
5. Glaucomatous damage sufficiently severe to prevent washout in the opinion of the examiner or visual field defect within 10 degrees of fixation
6. Glaucoma other than exfoliation syndrome
7. Absence of exfoliation material on the lens surface in the eye to be treated
8. Known allergy or sensitivity to any of the study medications
9. Ocular pathology that may interfere with the ability to obtain tonography, visual fields, or accurate IOP readings
10. Angle-closure glaucoma
11. Diabetic retinopathy
12. Previous intraocular or laser surgery.
13. Unwilling or unable to give consent
14. Pregnant or lactating women

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2000-08; Primary Completion 2007-09 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Latanoprost combined with pilocarpine (L-PILO) should be as effective as timolol or Cosopt in lowering IOP | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ritch, MD, Principal Investigator — New York Eye and Ear Infirmary
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States